CLINICAL TRIAL: NCT00241891
Title: Primary Care Obesity Prevention: One or Multiple Targets
Brief Title: Behavior Change Family Counseling to Reduce Rate of Weight Gain in At-Risk Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital of Philadelphia (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2005-7-4442; R01HL084056 (NIH)
Record Dates: First submitted 2005-10-17; First posted 2005-10-19 (Estimated); Last update posted 2015-04-07 (Estimated); Status verified 2015-04

CONDITIONS: Cardiovascular Diseases; Heart Diseases; Obesity
MeSH Terms: conditions — Cardiovascular Diseases; Heart Diseases; Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Healthy Lifestyle (Active Intervention) (Other): Parents and children in this program which will participate in a series of consultations and activities focused on multiple healthy interventions including healthy eating, drinking, and physical activity. The children will participate in a variety of age-appropriate games, activities and exercises that are focused on healthy eating, drinking, and physical activity. In addition, your child will receive information on developing healthy interpersonal and social skills.
  Interventions: Behavioral: Multiple behavior interventions
- Healthy Drinks (Active Intervention) (Other): Parents and children in this program will participate in a series of consultations and activities focused on a single intervention, the effects of beverage choices on diet, general health and teeth health. The children will participate in a variety of age-appropriate games, activities and exercises that are focused on beverages and health. In addition, your child will receive information on healthy nutrition, physical activity, and interpersonal and social skills.
  Interventions: Behavioral: Single behavior intervention
- Social and Leadership Skills (Control Intervention) (Other): Parents and children in this program will participate in a series of consultations that are designed to help your child learn strategies to make and keep friends, to express feelings appropriately, and to successfully decrease conflicts that often occur at school among children. The children will participate in a variety of age-appropriate games, activities and exercises that are focused on these friendship making strategies. In addition, your child will receive information on healthy nutrition and physical activity. There is o intervention with regards to healthy weight.
  Interventions: Behavioral: Control Intervention unrelated to weight

INTERVENTIONS:
Behavioral: Single behavior intervention — Focused on changing beverage choices which may have a significant impact on weight.
  Other Names: Focused on changing beverage choices with the goal
  Arms: Healthy Drinks (Active Intervention)
Behavioral: Multiple behavior interventions — Focused on multiple behaviors (nutrition, beverages, physical activity, and sedentary lifestyle) which may have a significant impact on weight.
  Arms: Healthy Lifestyle (Active Intervention)
Behavioral: Control Intervention unrelated to weight — Focused on standard intervention strategies unrelated to weight including bullying prevention.
  Arms: Social and Leadership Skills (Control Intervention)

SUMMARY:
This study will train primary care providers to counsel families on behavior change that is aimed at reducing the rate of weight gain in at-risk children.

DETAILED DESCRIPTION:
BACKGROUND:

In addition to family, school, and community, primary care is a promising setting for childhood obesity prevention. However, most pediatric primary care providers are not trained to deliver behavior modification interventions and, according to preliminary data, are less likely to address obesity prevention when they perceive insufficient time during well-care visits.

DESIGN NARRATIVE:

This is a controlled study of obesity prevention, with group randomization of two standardized 12-month intervention strategies at the practice level. The intervention strategies are based on the behavioral economics theory and will be delivered by primary care providers after training in behavior modification. The first strategy will target change in multiple behaviors, while the second strategy will target only one behavior (beverage consumption). These two interventions will be compared to an active control intervention that is unrelated to weight (bullying prevention). Six to seven primary care practices will be randomized to each arm with 21 patients per practice, for a total of 17 practices and 350 patients. The primary aim is to demonstrate that either obesity prevention intervention will result in less body mass index (BMI) increase (adjusted using z-score) in children age 8 to 12 years who are at risk for overweight (BMI 50th-95th percentile), as compared to a control intervention. The study also hypothesizes that the multiple-behavior intervention, the single-behavior intervention, or both will result in less adjusted BMI increase than the control intervention at 24 months post-randomization, with no a priori assumption in differences between the two obesity prevention strategies. Blood pressure, insulin resistance, dyslipidemia, and oral health status will be secondary outcomes. Intermediate behavioral outcomes and process data will be collected.

ELIGIBILITY:
Inclusion Criteria:

* Sought care at the participating practices at least once in the 3 years prior to study entry
* Children "at risk for overweight" at their last clinical visit (according to the Center for Disease Control and Prevention [CDC] definition of a BMI at or above the 50th percentile, but less than the 95th percentile)
* Children who consume at least 28 oz of sweetened beverages per week (i.e., an average of 4 oz per day) as assessed during the telephone screening by selected components of a validated food frequency questionnaire
* The following conditions will be acceptable if they have been well controlled in the 3 months prior to study entry: hypertension, dyslipidemia, sleep apnea, asthma, and insulin resistance without diabetes

Exclusion Criteria:

* Developmental delay requiring special education
* Depression
* Psychosis
* Eating disorder
* Significant orthopedic problems interfering with physical activity
* Diabetes
* Any significant chronic condition potentially interfering with nutrition or physical activity
* Treated with a drug known to affect weight gain
* Measured BMI z-score at first visit higher than +2.0 Standard Deviations (97.7th percentile)
* Families who are uninterested or unable to participate
* Home-schooled

Ages: 8 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 158 (Actual)
Dates: Start 2006-07; Primary Completion 2011-05 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
Changes in BMI z-score | Measured at Month 12

CONTACTS AND LOCATIONS:
Overall Officials: Stephen Leff, PhD, Principal Investigator — Children's Hospital of Philadelphia
Locations (1):
- The Children's Hospital of Philadelphia, Philadelphia, Pennsylvania, United States

REFERENCES:
- [Derived] Stettler N, Wrotniak BH, Hill DL, Kumanyika SK, Xanthopoulos MS, Nihtianova S, Shults J, Leff SS, Pinto A, Berkowitz RI, Faith MS. Prevention of excess weight gain in paediatric primary care: beverages only or multiple lifestyle factors. The Smart Step Study, a cluster-randomized clinical trial. Pediatr Obes. 2015 Aug;10(4):267-74. doi: 10.1111/ijpo.260. Epub 2014 Sep 24. PMID 25251166